CLINICAL TRIAL: NCT03922334
Title: Navigating New Motherhood 2: Patient Navigation to Improve Outcomes Among Low-income Women in the Postpartum Period
Brief Title: Navigating New Motherhood 2
Acronym: NNM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lynn M Yee, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU002096009; 1R01HD098178 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Health; Breastfeeding; Contraception; Preventive Care / Anticipatory Guidance; Retention in Care
MeSH Terms: conditions — Breast Feeding | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: There will be two cohorts: One cohort will be provided intensive, individualized, one-on-one navigation services through 12 weeks postpartum and, based on individual needs, ongoing, tapered navigation through one year (11-13 months) postpartum. The second cohort will receive usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation Group (Experimental): Women who are randomized into NNM2 will be assigned to a patient navigator. The patient navigator will meet with the patient during pregnancy and after delivery occurs for introductions and education. The patient navigator will offer support and resources (transportation, community referrals, support for your mental health, connection to your doctors, etc.). The navigator will also help to schedule postpartum medical appointments, and will remind the patients of these appointments via text, email, or phone calls. The navigator will continue to provide psychosocial support, social needs support, and continued linkage to resources through one-year postpartum.
  Interventions: Behavioral: Patient Navigation Program
- Non-navigation cohort (No Intervention): No navigation will be provided; women will receive usual care.

INTERVENTIONS:
Behavioral: Patient Navigation Program — A postpartum patient navigation program is designed to reduce barriers to care, enhance access, and improve multiple postpartum health outcomes, including retention in care, contraception uptake, vaccination, and depression screening.
  Arms: Navigation Group

SUMMARY:
The primary aim of this study is to determine whether implementation of a postpartum patient navigation program improves health outcomes among low-income women. Patient navigation is a barrier focused, long-term patient-centered intervention that offers support for a defined set of health services. The intervention under investigation is a comprehensive postpartum patient navigator program. Women who are randomized to receive patient navigation will be compared to women who are randomized to receive usual care. Navigators will support women through one year postpartum. The NNM2 program will be grounded in understanding and addressing social determinants of health in order to promote self-efficacy, enhance access, and sustain long-term engagement. Participants will undergo surveys, interviews, and medical record review at 4-12 weeks and 11-13 months postpartum. The investigators will additionally conduct focus groups and surveys with clinical providers.

DETAILED DESCRIPTION:
The postpartum period - often called the "fourth trimester" - is a time of rapid and intense change in the life of a woman and her family, and uptake of health care during this transition is critical to optimizing women's long-term health and the health of their subsequent pregnancies. The importance of postpartum care has been reinforced by professional organizations, yet postpartum care in the United States remains inadequate. Substantial racial/ethnic and socioeconomic disparities in health care uptake, quality, and outcomes exist. Improving health for all women requires the development of new, more comprehensive approaches to postpartum and interconceptional care. One potential model may be patient navigation, which is a barrier-focused, longitudinal, patient-centered intervention that offers support for a defined set of health services.

This protocol is to evaluate whether implementation of a postpartum patient navigation program improves health outcomes among low-income women. The investigators previously developed a postpartum patient navigation program, called Navigating New Motherhood (NNM), which introduced a clinic-level intervention in which a patient navigator assumed postpartum supportive and logistical responsibilities for low-income women. Navigation was associated with improvements in outcomes (retention in care, contraception uptake, vaccination, and depression screening) compared to those of a historical cohort. The investigators now propose to test the efficacy of the updated NNM model - called "NNM2" - via a randomized trial. The study will randomize 400 pregnant or postpartum women (1:1) with publicly-funded prenatal care to NNM2 versus usual care. Women randomized to navigation will be provided intensive, individualized, one-on-one navigation services through 12 weeks postpartum and, based on individual needs, ongoing, tapered navigation through one year postpartum. The NNM2 program will be grounded in understanding and addressing social determinants of health in order to promote self-efficacy, enhance access, and sustain long-term engagement. Participants will undergo surveys, interviews, and medical record review at 4-12 weeks and 11-13 months postpartum.

Aim 1 will evaluate whether the navigation program improves clinical outcomes at 4-12 weeks postpartum as measured via a composite of health status that includes retention in care, receipt of recommended counseling ("anticipatory guidance"), receipt of desired family planning method, postpartum depression screening/care, breastfeeding initiation/maintenance, and receipt of indicated vaccinations. Sub-Aims will include investigation of relevant outcomes at 11-13 months postpartum. Aim 2 will evaluate whether NNM2 improves patient-reported outcomes. Aim 3 additionally involves examining obstetric and primary care provider perspectives on the navigation program and on optimizing the postpartum transition. Completion of this study will fill an evidence gap by demonstrating whether postpartum patient navigation is an effective mechanism to improve women's short- and long-term health, enhance health care utilization, and improve patient and provider satisfaction.

NNM2 suspended enrollment due to COVID-19 beginning March 16, 2020. For already enrolled individuals, study visits and patient navigation activities were converted to tele-research and tele-navigation. Recruitment was planned to resume when the COVID-19 pandemic resolves and normal outpatient care has resumed. For individuals already recruited and whose care occurred during the early phases of the pandemic, the outcomes definitions were appropriately modified for the conduct of telemedicine during the pandemic. Recruitment resumed on June 8, 2020, with continued use of telemedicine or tele-research when appropriate. Given the ongoing pandemic, the modified outcomes definitions for telemedicine provision of care were retained.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (any plurality) delivering at or after 20 weeks of gestation OR postpartum (during hospitalization), regardless of perinatal outcome
* 16 years or older
* Low-income socioeconomic status (publicly funded prenatal care)
* Ability to speak and read English or Spanish
* Established patient at the Northwestern Medicine Prentice Ambulatory Care clinical site (at least one antenatal clinical visit).

Exclusion Criteria:

* Intent to transfer care to an outside institution
* HIV (as these patients already receive intensive social support and navigation-like services at this institution)
* Prior pregnancy in which individual declined participation
* Prior enrollment in NNM2
* Enrollment in a concurrent research study that poses a potential conflict to the aims of either NNM2 or the other study

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 405 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Postpartum health at 4-12 weeks after delivery | 4-12 weeks postpartum
  Number of women who achieve a composite measure of health status that includes retention in care, receipt of recommended counseling (anticipatory guidance), receipt of desired family planning method, postpartum depression screening and linkage, breastfeeding initiation and maintenance, and receipt of indicated vaccination. Components of the primary outcome composite will also be examined as a score and individually as secondary outcomes (see below). (Outcome is modified to include receipt telemedicine when appropriate for health care for women who require postpartum care during the pandemic)

SECONDARY OUTCOMES:
Retention in care (component of primary outcome) | 4-12 weeks postpartum
  Number of participants who return for comprehensive medical care at least once between 4 and 12 weeks postpartum.
Receipt of recommended counseling/anticipatory guidance (component of primary outcome) | 4-12 weeks and 1 year postpartum
  Number of participants who have been counseled about indicated topics recommended for postpartum care/health
Receipt of desired family planning method (component of primary outcome) | 4-12 weeks and 1 year postpartum
  Number of participants who received their desired family planning method
Postpartum depression screening and care (component of primary outcome) | 4-12 weeks and 1 year postpartum
  Number of participants who undergo appropriate screening for postpartum depression with either 1) screening that indicates no depressive symptoms, or 2) if depressive symptoms are identified, patient receives linkage to further care
Breastfeeding initiation and maintenance (component of primary outcome) | 4-12 weeks postpartum
  Number of participants who have initiated and maintained exclusive or partial breastfeeding
Receipt of indicated vaccinations (component of primary outcome) | 4-12 weeks postpartum
  Number of participants who received indicated vaccines (e.g. influenza, TDaP, HPV, MMR; based on individual need)
Postpartum diabetes screening | 4-12 weeks and 1 year postpartum
  Among women with gestational diabetes mellitus (GDM), number of women with completion of a 2-hour oral glucose tolerance test by 12 weeks postpartum and any other diabetes screening tests by 1 year postpartum
Postpartum atherosclerotic cardiovascular disease screening | 4-12 weeks and 1 year postpartum
  Overall and among women with ASCVD-associated adverse pregnancy outcomes, number of women who undergo indicated clinical assessments for blood pressure, lipids, weight, nutrition, activity
Gestational weight retention | 4-12 weeks and 1 year postpartum
  Difference between weight at delivery and 1) weight at early postpartum (4-12 weeks) and 2) weight at 1 year postpartum
Breastfeeding duration | 4-12 weeks and 1 year postpartum
  Total duration of exclusive or partial breastfeeding among women who initated breastfeeding
Postpartum transition to primary care | 1 year postpartum
  Number of women with appointment made and kept for primary care by 1 year postpartum
Patient-reported outcomes - self-efficacy, activation, engagement, quality of life, and other PROs | 4-12 weeks and 1 year postpartum
  Differences in self-efficacy, activation, quality of life, engagement, and other PROs between women who are randomized to navigation versus usual care, using the DHHS PROMIS and other validated measures of PROs.
  PROs to be measured include global health status (PROMIS Global Health), health literacy (Newest Vital Sign), depressive symptoms (Patient Health Questionnaire-9), pregnancy experience and pregnancy-related stress (Pregnancy Experience Scale - Brief, at 4-12 weeks only), patient activation (Patient Activation Measure), health-related self-efficacy (PROMIS Self-Efficacy - general), informational support (PROMIS Informational Support), perceived stress (Perceived Stress Scale), breastfeeding self-efficacy (Breastfeeding Self-Efficacy Scale), postpartum preparedness (Postpartum Preparedness Checklist), and satisfaction with prenatal and postpartum care (original and adaptation of Prenatal Care Satisfaction Scale).
Patient-reported outcomes - experiences with navigation (survey) | 4-12 weeks and 1 year postpartum
  Navigated participants' experiences with navigation as assessed through PRO surveys (Patient Satisfaction with Interpersonal Relationship with Navigator Scale and Patient Satisfaction with Logistical Aspects of Navigation Scale).
Experiences with navigation (qualitative) | 3-6 months postpartum and 1 year postpartum
  Qualitative perspectives on experiences with the navigation program, based on interviews with women who received navigation
Pregnancy/postpartum experiences during the pandemic | At any point during the COVID-19 pandemic, up to 3 months after the end of the pandemic
  Qualitative perspective of participants' experiences during the COVID-19 pandemic, utilizing a semi-structured interview guide developed by the research team, as it relates to their receipt of health care, experiences as a pregnant person and new parent, and the role of patient navigation in this time period

OTHER OUTCOMES:
Clinician perspectives on patient navigation | Through completion of study, an average of 3 years
  Qualitative feedback on how NNM2 can meet the needs of the clinicians and optimize postpartum care and the transition to primary care, as assessed by feedback from obstetrician and primary care provider focus groups
Clinician experiences with NNM2 | Through completion of study, an average of 5 years
  Number of clinicians who believed NNM2 met their needs and improved patient care, as determined by survey feedback obtained at the time of participants' postpartum visits
Navigation intensity and activities | Through completion of study, an average of 5 years
  Mixed methods data on navigation intensity (number of interactions over the postpartum year), types of activities completed for/with participants, types of communication modes used, and numbers/types of other health care team members involved in navigation activities. Data will be integrated from navigator weekly logs of navigation activities and quarterly in-depth qualitative interviews with the navigators.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Yee, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yee LM, Williams B, Green HM, Carmona-Barrera V, Diaz L, Davis K, Kominiarek MA, Feinglass J, Zera CA, Grobman WA. Bridging the postpartum gap: best practices for training of obstetrical patient navigators. Am J Obstet Gynecol. 2021 Aug;225(2):138-152. doi: 10.1016/j.ajog.2021.03.038. Epub 2021 Apr 1. PMID 33812809
- [Result] Ruderman RS, Dahl EC, Williams BR, Davis K, Feinglass JM, Grobman WA, Kominiarek MA, Yee LM. Provider Perspectives on Barriers and Facilitators to Postpartum Care for Low-Income Individuals. Womens Health Rep (New Rochelle). 2021 Jul 16;2(1):254-262. doi: 10.1089/whr.2021.0009. eCollection 2021. PMID 34318295
- [Result] Filicko A, Huennekens K, Davis K, Dolan BM, Williams BR, Feinglass J, Grobman WA, Kominiarek MA, Yee LM. Primary Care Clinician Perspectives on Patient Navigation to Improve Postpartum Care for Patients with Low Income. Womens Health Rep (New Rochelle). 2022 Dec 15;3(1):1006-1015. doi: 10.1089/whr.2022.0064. eCollection 2022. PMID 36636317
- [Result] Green HM, Diaz L, Carmona-Barrera V, Grobman WA, Yeh C, Williams B, Davis K, Kominiarek MA, Feinglass J, Zera C, Yee LM. Mapping the Postpartum Experience Through Obstetric Patient Navigation for Low-Income Individuals. J Womens Health (Larchmt). 2024 Jul;33(7):975-985. doi: 10.1089/jwh.2023.0459. Epub 2024 Jan 23. PMID 38265478
- [Result] Green HM, Carmona-Barrera V, Diaz L, Yeh C, Williams B, Davis K, Kominiarek MA, Feinglass J, Grobman WA, Zera C, Yee LM. Implementation of postpartum navigation for low-income individuals at an urban academic medical center. PLoS One. 2023 Feb 23;18(2):e0282048. doi: 10.1371/journal.pone.0282048. eCollection 2023. PMID 36821597
- [Result] Ruderman RS, Dahl EC, Williams BR, Feinglass JM, Kominiarek MA, Grobman WA, Yee LM. Obstetric Provider Perspectives on Postpartum Patient Navigation for Low-Income Patients. Health Educ Behav. 2023 Apr;50(2):260-267. doi: 10.1177/10901981211043117. Epub 2021 Oct 12. PMID 34636273
- [Derived] Green HM, Williams B, Diaz L, Carmona-Barrera V, Davis K, Feinglass J, Kominiarek MA, Dolan BM, Grobman WA, Yee LM. Evaluating feedback from an implementation advisory board to assess the rollout of a postpartum patient navigation program. Implement Sci Commun. 2024 May 3;5(1):50. doi: 10.1186/s43058-024-00589-6. PMID 38702751
- [Derived] Davis KM, Lu L, Williams B, Roas-Gomez MV, Leziak K, Jackson J, Feinglass J, Yee LM. The Stress of Parenting in the Postpartum Period During the COVID-19 Pandemic. Womens Health Rep (New Rochelle). 2022 Nov 9;3(1):895-903. doi: 10.1089/whr.2022.0029. eCollection 2022. PMID 36479375